CLINICAL TRIAL: NCT06480279
Title: Development of Artificial Intelligence Innovation for Assessing Fall Risk Using Clinical Neurological Studies With Transcranial Magnetic Stimulation and Quantitative Sensory Testing in the Thai Elderly
Brief Title: Assessing Fall Risk Using Transcranial Magnetic Stimulation and Quantitative Sensory Testing
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Collaborators: King Chulalongkorn Memorial Hospital (Other); National Research Council of Thailand (Other Government)
Responsible Party: Sponsor
Other Study IDs: COA No. 0607/2024
Record Dates: First submitted 2024-06-13; First posted 2024-06-28 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2024-06

CONDITIONS: Fall
Keywords: Transcranial Magnetic Stimulation; Quantitative Sensory Testing; Falls; Elderly

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Non-fallers: Elderly without history of fall
- Fallers-low risk: Elderly with a history of falling 1 time within the last year.
- Fallers-moderate risk: Elderly with a history of falling twice within the last year.
- Fallers-high risk: Elderly with a history of falling >2 times within the last year.

SUMMARY:
The elderly are at high risk of falls due to neurophysiological changes, such as motor and sensory impairment, that occur with aging. The incidence of falls in older adults is high, with approximately 30% of adults over the age of 65 falling at least once per year. Falls can lead to serious consequences such as fractures, hospitalization, and loss of independence. The changes in neurophysiology have also been found to decrease balance control in aging people, leading to postural instability. It is well-known that postural balance is influenced by sensory inputs, including touch, proprioception, vision, and vestibular, as well as motor output such as motor controls. Impairments in these systems contribute to postural instability and an increased risk of falling in the elderly.

DETAILED DESCRIPTION:
The data collection will be arranged in the same order. Practice trials will be provided before the start of the data collection. The entire data collection session will take approximately 90 minutes. Data collection will be conducted for both the baseline and the 3-month follow-up.

The data collection will include:

1. Demographic information such as age, sex, body height, body weight, body mass index, medical history, medical diagnosis, body composition, and the MoCA (Montreal Cognitive Assessment).
2. Neurophysiological assessments such as electromyography and Quantitative Sensory Testing (QST).
3. Functional tests such as the Timed up and go test and Chait stand test.

ELIGIBILITY:
Inclusion Criteria:

1) Male and female individuals aged 65-80 years.

Exclusion Criteria:

1. History of previous lower limb surgery, such as total knee replacement or ankle surgery.
2. History of a neurological disorder, such as stroke or Parkinson's disease.
3. History of vestibular disease, such as Meniere's disease.
4. History of seizures or epilepsy.
5. The presence of metal implanted devices in or around the head area
6. MoCA score < 26

Ages: 65 Years to 80 Years | Sex: All
Age Groups: Older Adult
Study Population: Thai elderly who have received check-ups or treatment at King Chulalongkorn Memorial Hospital, Bangkok, Thailand.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-08-16 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | MoCA will be measured at two time points (baseline and 3 months), through study completion, an average of 1 year.
  MoCa is a screening test used to detect mild cognitive decline and early signs of dementia. The total score of the test is 30 points.
  The MoCA will be recored in scores.
Body weight | Body weight will be measured at two time points (baseline and 3 months), through study completion, an average of 1 year.
  We will used the bioelectrical impedance analysis (BIA), which is a method used for measuring body composition.Participants will be asked to step on to the BIA device, placing their feet on the foot electrodes.
  The body weight will be recored in kilograms.
Muscle mass | Muscle mass will be measured at two time points (baseline and 3 months), through study completion, an average of 1 year.
  We will used the bioelectrical impedance analysis (BIA), which is a method used for measuring body composition.Participants will be asked to step on to the BIA device, placing their feet on the foot electrodes.
  The muscle mass will be recored in kilograms.
Body mass index (BMI) | BMI will be measured at two time points (baseline and 3 months), through study completion, an average of 1 year.
  We will used the bioelectrical impedance analysis (BIA), which is a method used for measuring body composition.Participants will be asked to step on to the BIA device, placing their feet on the foot electrodes.
  The BMI will be recored in kg/m^2.
Percent body fat | Percent body fat will be measured at two time points (baseline and 3 months), through study completion, an average of 1 year.
  We will used the bioelectrical impedance analysis (BIA), which is a method used for measuring body composition.Participants will be asked to step on to the BIA device, placing their feet on the foot electrodes.
  Percent body fat will be recored in percentage.
The duration during Timed Up and Go Test | TUG will be measured at two time points (baseline and 3 months), through study completion, an average of 1 year.
  The Timed Up and Go Test (TUG) is a test for assessing fall risk. Participants will begin by sitting on a chair. They will be asked to stand up, walk 3 meters away at a comfortable speed, turn around a traffic cone, walk back, and sit down.
  TUG will be recored in second.
The repetition of Chair Stand Test | Chair Stand Test will be measured at two time points (baseline and 3 months), through study completion, an average of 1 year.
  Chair Stand Test is used to test leg strength and endurance. Participants will begin by sitting on a chair. Participants will be instructed to stand up with full leg extension as quickly as possible, sit back down as quickly as possible, andrepeat this process for 30 seconds.
  Chair Stand Test will be recorded in repetition.
Muscle evoke potential (MEP) | Muscle evoke potential will be measured at two time points (baseline and 3 months), through study completion, an average of 1 year.
  Participants will be stimulated at the primary motor cortex by transcranial magnetic stimulation to measure cortical excitability, which sends the motor outputs to Tibialis Anterior (TA) and Abductor Pollicis Brevis (APB) muscles. The MEP will be used to assess muscle activity in these muscles during the stimulation.
  The MEP will be measured in mV.
Cortical silent period (CSP) | Muscle evoke potential will be measured at two time points (baseline and 3 months), through study completion, an average of 1 year.
  Participants will be stimulated at the primary motor cortex by transcranial magnetic stimulation to measure cortical excitability, which sends the motor outputs to Tibialis Anterior (TA) and Abductor Pollicis Brevis (APB) muscles. The CSP will be used to assess muscle activity in these muscles during the stimulation.
  The CSP will be measured in ms.
Cold temperature threshold | Cold temperature threshold will be measured at two time points (baseline and 3 months), through study completion, an average of 1 year.
  Participants will be stimulated by Quantitative Sensory Testing (QST) with cold temperature on their legs. QST is the standard device validated by the manufacturer and approved for use in research assessments, as demonstrated in the supplementary files.
  Cold temperature threshold will be measure in degree Celsius.
Vibration threshold | Vibration temperature threshold will be measured at two time points (baseline and 3 months), through study completion, an average of 1 year.
  Participants will be stimulated by Quantitative Sensory Testing (QST) with vibration threshold on their legs. QST is the standard device validated by the manufacturer and approved for use in research assessments, as demonstrated in the supplementary files.
  Vibration threshold will be measure in μm.

CONTACTS AND LOCATIONS:
Overall Officials: Jakkrit Amornvit, MD, Principal Investigator — Chulalongkorn University; Phunsuk Kantha, PT.,PhD, Principal Investigator — Mahidol University; Kulvara Lapanan, PT, Principal Investigator — Chulalongkorn University
Locations (1):
- Department of Medicine, Faculty of Medicine, Chulalongkorn University., Bangkok, Thailand